CLINICAL TRIAL: NCT06359665
Title: A Randomized Controlled Trial of Oral Curcumin for the Treatment of Pain of CMC Arthritis
Brief Title: Oral Curcumin for the Treatment of Pain of Thumb Base Joint (CMC) Arthritis
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Brent DeGeorge (Other)
Responsible Party: Sponsor-Investigator, Brent DeGeorge, Associate Professor of Plastic Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSR230544
Record Dates: First submitted 2024-03-15; First posted 2024-04-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Arthritis of Carpometacarpal Joint of Left Thumb; Arthritis of Carpometacarpal Joint of Right Thumb
Keywords: Thumb carpometacarpal osteoarthritis (CMC OA); Thumb carpometacarpal Osteoarthritis; turmeric; curcumin
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: The study design will be a double-blind, randomized controlled trial with crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral curcumin (Experimental): Oral curcumin 500 mg capsules taken twice each day for 4 weeks.
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): Oral placebo capsules taken twice each day for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcumin — 500 mg capsule twice daily
  Other Names: Nature Made, PharmaVite LLC; Turmeric
  Arms: Oral curcumin
Drug: Placebo — capsule twice daily
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the use of turmeric (Curcumin) as a treatment for pain of thumb-joint arthritis. Turmeric is commonly being used as an over-the-counter treatment for musculoskeletal pain. Clinical trials have demonstrated a pain-relief benefit for knee osteoarthritis, however no clinical trial has been performed to establish efficacy of curcumin in humans for thumb-joint arthritis. The main question[s] it aims to answer are:

* Is Turmeric more effective than placebo at relieving pain for thumb-joint arthritis? A placebo is a look-alike substance that contains no active drug.
* Is Turmeric more effective than placebo at improving patient-reported outcomes for CMC arthritis?
* Is Turmeric safe for participants with thumb-joint arthritis?

Participants will:

* take 4 weeks of daily Turmeric capsules,
* take 4 weeks of daily placebo capsules
* answer daily surveys about how they are feeling and functioning.

DETAILED DESCRIPTION:
This randomized controlled trial of oral curcumin for the treatment of pain of CMC arthritis will investigate the therapeutic potential of curcumin as an oral treatment for pain of CMC arthritis. Rationale: Curcumin is commonly being used as an over-the-counter treatment for musculoskeletal pain. Clinical trials have demonstrated a pain-relief benefit for knee osteoarthritis, however no clinical trial has been performed to establish efficacy of curcumin in humans for CMC arthritis. Hypothesis: Curcumin is more effective than placebo for relieving pain and improving patient-reported outcomes for CMC arthritis Study Design: The study design will be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 4 weeks of the Curcumin or control and then crossover to the other condition for 4 additional weeks. Patients will take the oral curcumin or control placebo capsule twice daily. Subjects will be advised to observe adverse effects.

The study design will be a double-blind randomized control trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 4 weeks of the case (curcumin) or control capsules and then crossover to the other condition for 4 more weeks with a 2-week washout interval between. Patients will take one oral capsule by mouth twice daily. The subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects. If mild to severe adverse events are noticed, the patient's will discontinue the use of the capsules, and appropriate care and observation will be taken. Each condition will last for 4 weeks and then subjects will be contacted by the study coordinator to facilitate crossover into the other condition following a 2-week washout period. To capture any delayed-onset adverse events, subjects will attend a follow-up visit seven days following the last dose of the curcumin capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 years or older.
4. For females, must be willing to use an approved form of birth control during this study. Acceptable forms of birth control:

   * Norplant
   * IUD (intrauterine device)
   * Birth Control Patch
   * Depo-Provera
   * Sterilization

   The following may be used if combined with other birth control methods:
   * Condoms
   * Diaphragm
   * Jellies or foam
   * Cervical cap
   * Sponge
5. For males, must be willing to not father a baby for the duration of the study and for 90 days after the last dose of study drug, or donate to a sperm back during this time. Must be willing to use an approved form of birth control during this time. Acceptable forms of birth control:

   * Condoms
   * Sterilization
6. Daily visual analog pain greater than 5 and ≤ 9 out of 10.
7. Duration of pain for greater than 30 days.
8. Presence of radiographically confirmed diagnosis of thumb basal joint arthritis

Exclusion Criteria:

1. Participant does not speak English.
2. Participant is blind.
3. Severe cardiac, pulmonary, liver, gastrointestinal and hematological disease (including coagulopathy), and /or renal disease.
4. Abnormal hematological, coagulation, and/or liver function test results.
5. Coumadin use at time of screening.
6. Use of any anticoagulant and antiplatelet medication.
7. History of mental illness.
8. Participant who is incarcerated.
9. History of drug or substance abuse.
10. Pre-existing curcumin or turmeric product usage within 3 months of the study period.
11. Participant has had a corticosteroid injection ≤ 60 days prior.
12. Participant has had prior surgery for osteoarthritis treatment
13. Participant who has fibromyalgia and post-operative pain.
14. Females who are pregnant, nursing or planning a pregnancy
15. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates of CYP3A4:

    * Itraconazole,
    * Ketoconazole,
    * Azamulin,
    * Troleandomycin,
    * Verapamil,
    * John's wart,
    * Phenobarbital,
16. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates of CYP2C19:

    * Nootkatone,
    * Ticlopidine,
    * Rifampin,
    * Omeprazole),
17. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates of CYP2C8:

    * Montelukast,
    * Quercetin,
    * Phenelzine,
    * Rifampin,
    * Clopidogrel ,
18. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates of CYP2C9:

    * Sulfaphenazole,
    * Tienilic acid,
    * Carbamazepine,
    * Apoflutamide ,
    * Fluconazole,
    * Celecoxib,
19. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates of CYP1A2:

    * alpha-Naphthoflavone,
    * Furafylline,
    * Phenytoin,
    * Rifampin,
    * Ritonavir,
    * smoking,
    * Teriflunomide,
    * Ciprofloxacin,
    * oral contraceptives,
    * Allopurinol
20. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates of CYP2B6 :

    * Sertraline,
    * Phencyclidine,
    * Thiotepa,
    * Ticlopidine,
    * Carbamazepine,
    * Efavirenz,
    * Rifampin,
    * Bupropion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain on the Visual Analog Pain (VAS) Score | Baseline and Week 4, Week 6
  The Visual Analog Pain (VAS) Score is a validated, self-reported subjective measure for measuring acute and chronic pain. Possible scores range from 0 (no pain) to 10 (worst possible pain). Change = (Week (4 or 6) Score - Baseline Score).a validated, self-report
Change from Baseline in Pain on the Visual Analog Pain (VAS) Score - crossover condition | Baseline and Week 10, Week 12
  The Visual Analog Pain (VAS) Score is a validated, self-reported subjective measure for measuring acute and chronic pain. Possible scores range from 0 (no pain) to 10 (worst possible pain). Change = (Week Change = (Week (10 or 12) Score - Baseline Score).

SECONDARY OUTCOMES:
Change from Baseline in Normal Function on the Single Assessment Numerical Evaluation (SANE) Score | Baseline and Week 4, Week 6
  The SANE Score is a self-reported subjective measure for measuring percentage of normal function. Possible scores range from 0 (most abnormal) to 100 (normal). Change = (Week (4 or 6) Score - Baseline Score)
Change from Baseline in Normal Function on the Single Assessment Numerical Evaluation (SANE) Score - crossover condition | Baseline and Week 10, Week 12
  The SANE Score is a self-reported subjective measure for measuring percentage of normal function. Possible scores range from 0 (most abnormal) to 100 (normal). Change = (Week 10, Week 12 Score - Baseline Score)
Change from Baseline in Quality of Life on the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health-10 Score | Baseline and Week 4, Week 6
  The PROMIS Global Health-10 is a validated, self-reported subjective measure for measuring generic health related quality of life. Possible scores range from 0 (most severe impairment) to 20 (best health). Change = (Week (4 or 6) Score - Baseline Score)
Change from Baseline in Quality of Life on the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health-10 Score - crossover condition | Baseline and Week 10, Week 12
  The PROMIS Global Health-10 is a validated, self-reported subjective measure for measuring generic health related quality of life. Possible scores range from 0 (most severe impairment) to 20 (best health). Change = (Week (10 or 12) Score - Baseline Score)
Change from Baseline in Pain interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score | Baseline and Week 4, Week 6
  The PROMIS Pain Interference is a validated, self-reported subjective measure for measuring generic health related quality of life. Possible scores range from 0 (does not interfere) to 10 (completely interferes). Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in Pain interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score - crossover condition | Baseline and Week 10, Week 12
  The PROMIS Pain Interference is a validated, self-reported subjective measure for measuring generic health related quality of life. Possible scores range from 0 (does not interfere) to 10 (completely interferes). Change = (Week (10, 12) Score - Baseline Score)
Change from Baseline in Pain interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Upper Extremity (UE) Score | Baseline and Week 4, Week 6
  The PROMIS UE computer adaptive test is a validated computer adaptive test to assess upper extremity functional status. Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in Pain interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Upper Extremity (UE) Score | Baseline and Week 10, Week 12
  The PROMIS UE computer adaptive test is a validated computer adaptive test to assess upper extremity functional status. Change = (Week (10, 12) Score - Baseline Score)
Change from Baseline in Pain on the Australian/Canadian Hand Osteoarthritis (AUSCAN) Index | Baseline and Week 4, Week 6
  The AUSCAN Index is a 15-item scale measuring pain (5 items), stiffness (1 item) and function (9 items) during the preceding 48 hours. Possible scores range from 0 (none) to 4 (extreme). Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in Pain on the Australian/Canadian Hand Osteoarthritis (AUSCAN) Index | Baseline and Week 10, Week 12
  The AUSCAN Index is a 15-item scale measuring pain (5 items), stiffness (1 item) and function (9 items) during the preceding 48 hours. Possible scores range from 0 (none) to 4 (extreme). Change = (Week (10, 12) Score - Baseline Score)
Change from Baseline in Disability on The Quick Disability of the Arm, Shoulder (QuickDASH). | Baseline and Week 4
  The QuickDASH is a validated, self-reported 11-item scale measuring disability. Possible scores range from 0 (no disability) to 100 (most severe disability. Change = (Week 4 Score - Baseline Score)
Change from Baseline in Disability on The Quick Disability of the Arm, Shoulder (QuickDASH) - crossover condition | Baseline and Week 10
  The QuickDASH is a validated, self-reported 11-item scale measuring disability. Possible scores range from 0 (no disability) to 100 (most severe disability. Change = (Week 10 Score - Baseline Score)
Change from Baseline in perseverance on the Brief Resilience Index (BRI) | Baseline and Week 4, Week 6
  The BRI is a validated, self-reported 6-item validated tool to assess for resilience. Possible scores range from 1 (low resilience) to 5 (high resilience). Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in perseverance on the Brief Resilience Index (BRI) - crossover condition | Baseline and Week 10, Week 12
  The BRI is a validated, self-reported 6-item validated tool to assess for resilience. Possible scores range from 1 (low resilience) to 5 (high resilience). Change = (Week (10, 12) Score - Baseline Score)
Number of Participants With Treatment-Related Adverse Events | Through study completion, an average of 12 weeks
  Treatment-related adverse events will be reported throughout the study by self-report and clinician-driven questions at each visit
Change from Baseline in the Mean Seated Trough Cuff Systolic Blood Pressure | Baseline and Week 4
  Blood pressure (SBP and DBP) in mmHg using Sphygmomanometer will be assessed by the researchers at baseline and follow-up
Change from Baseline in heart rate | Baseline and Week 4
  Heartbeats per minute (BPM) will be assessed by the researchers at baseline and follow-up
Change from Baseline in the Mean Seated Trough Cuff Systolic Blood Pressure | Week 4 and Week 6
  Blood pressure (SBP and DBP) in mmHg using Sphygmomanometer will be assessed by the researchers at baseline and follow-up
Change from Baseline in heart rate | Week 4 and Week 6
  Heartbeats per minute (BPM) will be assessed by the researchers at baseline and follow-up
Change from baseline in serum liver panel parameters: Alanine transaminase (ALT), Alkaline phosphatase (ALP) and Aspartate aminotransferase (AST) | Through study completion, an average of 12 weeks
  Change from baseline in serum liver panel parameters: ALT, ALP and AST (International units per liter) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: glucose, blood urea nitrogen (BUN), Creatinine, Calcium | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: glucose, BUN, Creatinine, Calcium (mg/dL) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: estimated glomerular filtration rate (eGFR) | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: eGFR (mL/min/1.73m2) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Bilirubin | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Bilirubin (umol/L) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Sodium, Potassium, Chloride, Carbon Dioxide | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Sodium, Potassium, Chloride, Carbon Dioxide (meq/L) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Protein, Albumin | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Protein, Albumin (g/dL) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Prothrombin time- International normalized ratio (PT-INR) | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Prothrombin time- International normalized ratio (PT (seconds)-INR) at baseline and follow up
Change from baseline in serum complete blood count (CBC) parameters: Red Blood Cells (CBC), White Blood Cells (WBC), Platelets | Through study completion, an average of 12 weeks
  Change from baseline in serum complete blood count (CBC) parameters: RBC, WBC, Platelets (uL) at baseline and follow up
Change from baseline in serum complete blood count (CBC) parameters: Hemoglobin | Through study completion, an average of 12 weeks
  Change from baseline in serum complete blood count (CBC) parameters: Hemoglobin (g.dL) at baseline and follow up
Change from baseline in serum complete blood count (CBC) parameters: Hematocrit | Through study completion, an average of 12 weeks
  Change from baseline in serum complete blood count (CBC) parameters: Hematocrit (percentage) at baseline and follow up
Change from baseline in serum complete blood count (CBC) parameters: Mean Corpuscular Volume (MCV) | Through study completion, an average of 12 weeks
  Change from baseline in serum complete blood count (CBC) parameters: Mean Corpuscular Volume (MCV) (pg) at baseline and follow up
Change from baseline in serum complete blood count (CBC) parameters: the amount of hemoglobin per red blood cell.(MCH) | Through study completion, an average of 12 weeks
  Change from baseline in serum complete blood count (CBC) parameters: the amount of hemoglobin per red blood cell.(MCH) (pg) at baseline and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Brent DeGeorge, MD, PhD, Principal Investigator — University of Virginia Department of Plastic Surgery
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolf JM, Atroshi I, Zhou C, Karlsson J, Englund M. Sick Leave After Surgery for Thumb Carpometacarpal Osteoarthritis: A Population-Based Study. J Hand Surg Am. 2018 May;43(5):439-447. doi: 10.1016/j.jhsa.2017.11.019. Epub 2018 Feb 7. PMID 29428245
- [Background] Brat GA, Agniel D, Beam A, Yorkgitis B, Bicket M, Homer M, Fox KP, Knecht DB, McMahill-Walraven CN, Palmer N, Kohane I. Postsurgical prescriptions for opioid naive patients and association with overdose and misuse: retrospective cohort study. BMJ. 2018 Jan 17;360:j5790. doi: 10.1136/bmj.j5790. PMID 29343479
- [Background] Funk JL, Frye JB, Oyarzo JN, Kuscuoglu N, Wilson J, McCaffrey G, Stafford G, Chen G, Lantz RC, Jolad SD, Solyom AM, Kiela PR, Timmermann BN. Efficacy and mechanism of action of turmeric supplements in the treatment of experimental arthritis. Arthritis Rheum. 2006 Nov;54(11):3452-64. doi: 10.1002/art.22180. PMID 17075840
- [Background] Lakhan SE, Ford CT, Tepper D. Zingiberaceae extracts for pain: a systematic review and meta-analysis. Nutr J. 2015 May 14;14:50. doi: 10.1186/s12937-015-0038-8. PMID 25972154
- [Background] Goel A, Kunnumakkara AB, Aggarwal BB. Curcumin as "Curecumin": from kitchen to clinic. Biochem Pharmacol. 2008 Feb 15;75(4):787-809. doi: 10.1016/j.bcp.2007.08.016. Epub 2007 Aug 19. PMID 17900536
- [Background] Daily JW, Yang M, Park S. Efficacy of Turmeric Extracts and Curcumin for Alleviating the Symptoms of Joint Arthritis: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. J Med Food. 2016 Aug;19(8):717-29. doi: 10.1089/jmf.2016.3705. PMID 27533649
- [Background] Travica N, Teasdale S, Marx W. Nutraceuticals in mood disorders: current knowledge and future directions. Curr Opin Psychiatry. 2023 Jan 1;36(1):54-59. doi: 10.1097/YCO.0000000000000826. Epub 2022 Aug 29. PMID 36044293
- [Background] Hafez Ghoran S, Calcaterra A, Abbasi M, Taktaz F, Nieselt K, Babaei E. Curcumin-Based Nanoformulations: A Promising Adjuvant towards Cancer Treatment. Molecules. 2022 Aug 16;27(16):5236. doi: 10.3390/molecules27165236. PMID 36014474
- [Background] Zeng L, Yang T, Yang K, Yu G, Li J, Xiang W, Chen H. Efficacy and Safety of Curcumin and Curcuma longa Extract in the Treatment of Arthritis: A Systematic Review and Meta-Analysis of Randomized Controlled Trial. Front Immunol. 2022 Jul 22;13:891822. doi: 10.3389/fimmu.2022.891822. eCollection 2022. PMID 35935936
- [Background] Bannuru RR, Osani MC, Al-Eid F, Wang C. Efficacy of curcumin and Boswellia for knee osteoarthritis: Systematic review and meta-analysis. Semin Arthritis Rheum. 2018 Dec;48(3):416-429. doi: 10.1016/j.semarthrit.2018.03.001. Epub 2018 Mar 10. PMID 29622343
- [Background] Hsiao AF, Lien YC, Tzeng IS, Liu CT, Chou SH, Horng YS. The efficacy of high- and low-dose curcumin in knee osteoarthritis: A systematic review and meta-analysis. Complement Ther Med. 2021 Dec;63:102775. doi: 10.1016/j.ctim.2021.102775. Epub 2021 Sep 16. PMID 34537344
- [Background] Wang Z, Singh A, Jones G, Winzenberg T, Ding C, Chopra A, Das S, Danda D, Laslett L, Antony B. Efficacy and Safety of Turmeric Extracts for the Treatment of Knee Osteoarthritis: a Systematic Review and Meta-analysis of Randomised Controlled Trials. Curr Rheumatol Rep. 2021 Jan 28;23(2):11. doi: 10.1007/s11926-020-00975-8. PMID 33511486
- [Background] Kuptniratsaikul V, Dajpratham P, Taechaarpornkul W, Buntragulpoontawee M, Lukkanapichonchut P, Chootip C, Saengsuwan J, Tantayakom K, Laongpech S. Efficacy and safety of Curcuma domestica extracts compared with ibuprofen in patients with knee osteoarthritis: a multicenter study. Clin Interv Aging. 2014 Mar 20;9:451-8. doi: 10.2147/CIA.S58535. eCollection 2014. PMID 24672232

DOCUMENTS (1):
  • Informed Consent Form (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT06359665/ICF_000.pdf